CLINICAL TRIAL: NCT05960110
Title: Randomized Clinical Trial to Evaluate the Impact on Oral Health of the "Oral Health Package Law" (School Daily Brushing Program) Combined, or Not, With Fluor Varnish Application on Schoolchildren of Mérida, Mexico.
Brief Title: Randomized Clinical Trial: Oral Health Package Law and Fluor Varnish Impact on Schoolchildren in Merida, Mexico
Acronym: DBMX
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Anahuac Mayab University (Other)
Collaborators: Colgate Palmolive (Industry)
Responsible Party: Principal Investigator, Mildred Beatriz Salas Ley, DDS orthodontic specialist, Anahuac Mayab University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AnahuacMayabU; EXT-2023-02-DB-FV-MEX (Other: Anahuac Mayab University)
Record Dates: First submitted 2023-07-18; First posted 2023-07-25 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Caries; Gum Disease
Keywords: Caries, gum disease
MeSH Terms: conditions — Gingival Diseases

STUDY DESIGN:
Intervention Model Description: A parallel randomized single-blinded clinical trial
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor will be blinded to the treatment allocation of the participants. Coded data sheets are used to maintain the blinding
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Group (Experimental): Fluoride toothpaste and fluoride varnish
  Interventions: Drug: Fluoride varnish
- Control Group (Sham Comparator): Fluoride toothpaste
  Interventions: Drug: Fluoride toothpaste

INTERVENTIONS:
Drug: Fluoride varnish — Fluoride varnish 26200 ppm
  Arms: Test Group
Drug: Fluoride toothpaste — Fluoride toothpaste 1450 ppm
  Arms: Control Group

SUMMARY:
Study aimed at evaluating the impact on oral health of the "Ley del Paquete de Salud Bucal" (daily school brushing program) combined, or not, with the application of fluoride varnish in schoolchildren from 6 to 8 years old who attend public elementary schools in Mérida,

Mexico. with a two-year follow-up (2023-2025).

DETAILED DESCRIPTION:
First visit:

The child will be asked to report to the school clinic to be screened by the dentist and/or hygienist to determine if he or she is a suitable test subject. If the parents and the child decide to participate and is accepted into the study, the family need to follow a specific set of instructions. The child will not perform or receive any oral hygiene (other than that described below).

At the beginning of the study, the child's teeth and gums will be examined to determine if they are eligible to participate in the study. The parents/tutors will agree to use only the fluoride toothpaste provided for the duration of the study and will be required to brush

their teeth daily in the school setting. There will be no restrictions regarding eating habits. A clinical score will be made to assess the level of caries, gingivitis and plaque level of all teeth and will be recorded on the evaluation forms. Questionnaires will be completed, and the child will be provided with a medium soft-bristled toothbrush and a tube of household toothpaste. Supervised brushing will be performed by asking the child to coat the

toothbrush head with their assigned toothpaste and brush their teeth for two (2) minutes. Subsequently, the child may receive a topical application of fluoride varnish depending on which group they belong to in this clinical trial.

The participants and their family will be asked if they want to participate in the

teleconsultation program where they will have access to an information platform with sessions to connect with a professional to obtain oral health guidance.

Teleconsultation control - 3 months (optional)

They will be able to schedule a teleconsultation visit where they will connect with a dental professional to receive individualized care and recommendations for the child's oral health.

Visit 2 (6 months)

At the 6-month visit, the child's teeth and gums will be examined. They will agree to use only the fluoride toothpaste provided to them for the duration of the study and will be required to brush their teeth daily in the school setting. There will be no restrictions

regarding eating habits.

A clinical score will be made to assess the level of caries, gingivitis and plaque level of all teeth and will be recorded on the evaluation forms. Questionnaires will be completed and the child will be provided with a medium soft-bristled toothbrush and a tube of household toothpaste. Supervised brushing will be performed by asking the child to coat the

toothbrush head with their assigned toothpaste and brush their teeth for two (2) minutes. Subsequently, the child may receive a topical application of fluoride varnish depending on which group they belong to in this clinical trial.

Teleconsultation control - 9 months (optional)

They will be able to schedule a teleconsultation visit where they will connect with a dental professional to receive individualized care and recommendations for the child's oral health.

Visit 3 (12 months)

At the 12-month visit, the child's teeth and gums will be examined. They will agree to use only the fluoride toothpaste provided to them for the duration of the study and will be

required to brush their teeth daily in the school setting. There will be no restrictions regarding eating habits.

A clinical score will be made to assess the level of caries, gingivitis and plaque level of all teeth and will be recorded on the evaluation forms. Questionnaires will be completed and the child will be provided with a medium soft-bristled toothbrush and a tube of household toothpaste. Supervised brushing will be performed by asking the child to coat the

toothbrush head with their assigned toothpaste and brush their teeth for two (2) minutes. Subsequently, the child may receive a topical application of fluoride varnish depending on which group they belong to in this clinical trial.

Consultation control - 15 months (optional)

They will be able to schedule a teleconsultation visit where they will connect with a dental professional to receive individualized care and recommendations for the child's oral health.

Visit 4 (18 months)

At the 18-month visit, the child's teeth and gums will be examined. They will agree to use only the fluoride toothpaste provided to them for the duration of the study and will be

required to brush their teeth daily in the school setting. There will be no restrictions regarding eating habits.

A clinical score will be made to assess the level of caries, gingivitis and plaque level of all teeth and will be recorded on the evaluation forms. Questionnaires will be completed and the child will be provided with a medium soft-bristled toothbrush and a tube of household toothpaste. Supervised brushing will be performed by asking the child to coat the

toothbrush head with their assigned toothpaste and brush their teeth for two (2) minutes. Subsequently, the child may receive a topical application of fluoride varnish depending on which group they belong to in this clinical trial.

Consultation control - 21 months (optional)

They will be able to schedule a teleconsultation visit where they will connect with a dental professional to receive individualized care and recommendations for the child's oral health.

Visit 5 (24 months)

At the 24-month visit, the child's teeth and gums will be examined. They will agree to use only the fluoride toothpaste provided to them for the duration of the study and will be

required to brush their teeth daily in the school setting. There will be no restrictions regarding eating habits.

A clinical score will be made to assess the level of caries, gingivitis and plaque level of all teeth and will be recorded on the evaluation forms. Questionnaires will be completed and the child will be provided with a medium soft-bristled toothbrush and a tube of household toothpaste. Supervised brushing will be performed by asking the child to coat the

toothbrush head with their assigned toothpaste and brush their teeth for two (2) minutes. Subsequently, the child may receive a topical application of fluoride varnish depending on which group they belong to in this clinical trial.

While participating as a subject in this study, the child may not use any oral product other than the one given to him. The child cannot participate as a subject in any other clinical study. Also, the child may not use drugs, except over-the-counter pain relievers, during the course of the study. The parents or legal guardians agree to inform the investigator of any new medications the child plans to take, including, but not limited to, antibiotics, antiseptics, decongestants, and antihistamines.

ELIGIBILITY:
Inclusion Criteria:

* 1. Men and women, between 6-8 years of age;
* 2. Children enrolled in first, second and third grade of primary education
* 3. Availability during the duration of the study;
* 4. Good general health (absence of any condition that, in the opinion of the Principal Investigator, could constitute a risk to the subject while participating in the study.
* 5 Examples include heart problems, valve/hip replacements, etc.);
* 6 Willingness to provide information related to his medical history;
* 7 Informed consent form signed by the caregiver;
* 8 Informed consent signed by the child

Exclusion Criteria:

* 1 Subjects must not have any of the following:
* 2 The caregiver is unwilling to sign the informed consent form
* 3 Subject participating in any other clinical study;
* 4. Subject allergic to oral care products, consumer personal care products or their ingredients;
* 5. Subjects with orthodontic bands, removable partial dentures, tumors of the hard parts or soft tissue of the oral cavity, or advanced periodontal disease
* 6. Continued use of medications known to affect gingival tissues (ie, calcium channel blockers, phenytoin, cyclosporine);
* 7. Subject is currently receiving chemotherapy
* 8. Subject has leukemia

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 900 (Estimated)
Dates: Start 2023-06-22 (Actual); Primary Completion 2025-12-22 (Estimated); Study Completion 2026-02-22 (Estimated)

PRIMARY OUTCOMES:
Impact on oral health | 24 months
  To evaluate the impact on oral health of the "Ley del Paquete de Salud Bucal" (daily school brushing program) combined, or not, with the application of fluoride varnish in schoolchildren from 6 to 8 years old who attend public elementary schools in Mérida, Mexico.

SECONDARY OUTCOMES:
Caries assessment | 24 months
  Caries will be evaluated by International Caries Detection and Assessment System (ICDAS) score
Gingivitis assessment | 24 months
  Gingivitis will be evaluated by Silness-Löe Index
Plaque assessment | 24 months
  Plaque assessment will be evaluated by Silness-Löe Index

CONTACTS AND LOCATIONS:
Locations (1):
- Anahuac Mayab University, Mérida, Yucatán, Mexico

IPD SHARING:
Plan to Share IPD: No